CLINICAL TRIAL: NCT03314467
Title: Role of Obstructive Sleep Apnea Syndrome in the Occurrence of Diabetic Retinopathy in Type 2 Diabetes.
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Principal Investigator, Marie Bruyneel, Chef de clinique, Centre Hospitalier Universitaire Saint Pierre
Other Study IDs: BE76201733442
Record Dates: First submitted 2017-10-16; First posted 2017-10-19 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Diabetes Mellitus; Obstructive Sleep Apnea
Keywords: diabetic retinopathy; diabetes; arterial hypertension; obstructive sleep apnea syndrome
MeSH Terms: conditions — Diabetes Mellitus; Sleep Apnea, Obstructive; Diabetic Retinopathy; Hypertension | interventions — Polysomnography; Arterial Pressure; Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — bloodserum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cases DR: diabetic patients with diabetic retinopathy (DR)
  Interventions: Diagnostic Test: polysomnography
- Cases other: diabetic patiens with other/multiple ocular disorder(s)
  Interventions: Diagnostic Test: polysomnography
- Control: diabetic patients without ocular abnormalities
  Interventions: Diagnostic Test: polysomnography

INTERVENTIONS:
Diagnostic Test: polysomnography — * classical polysomnography
  * non invasive measurement of blood pressure
  * blood test: determination of HbA1c, glucose, C-peptide, hemoglobin, white blood cell count, trombocytes
  Other Names: arterial tension; blood test

SUMMARY:
Diabetic retinopathy (DR) is the most common visual complication of diabetes. Risk factors for developing DR are diabetes duration, glycemic control, and hypertension . The prevalence ranges from 17 to 61% according to the diabetes duration .

Obstructive sleep apnea syndrome (OSAS) is very frequent in Type 2 Diabetes population, reaching a prevalence of 23-48% .

Few is known about the exact role of OSAS in the development of DR. A recent study has shown that OSAS is an independent predictor for the progression to pre-/proliferative DR. The purpose of the present study is to assess if the presence of OSA in diabetic patients is a predictive factor for DR occurrence.

DETAILED DESCRIPTION:
Diabetic retinopathy (DR) is the most common visual complication of diabetes. Risk factors for developing DR are diabetes duration, glycemic control, and hypertension. The prevalence ranges from 17 to 61% according to the diabetes duration.

Obstructive sleep apnea syndrome (OSAS) is very frequent in Type 2 Diabetes population, reaching a prevalence of 23-48%.

Few is known about the exact role of OSAS in the development of DR. A recent study has shown that OSAS is an independent predictor for the progression to pre-/proliferative DR. The purpose of the present study is to assess if the presence of OSA in diabetic patients is a predictive factor for DR occurrence.

ELIGIBILITY:
Inclusion Criteria:

* presence of diabetic type II
* able to undergo an in-lab polysomnography

Exclusion Criteria:

* known presence of obstructive sleep apnea and treated by CPAP

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a diagnosis of diabetes type I or type II who went to a ocular screening visit to assess ocular complications associated with diabetes are asked to undergo an in-lab polysomnography..
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Presence of obstructive sleep apnea in diabetic patients is a predictive factor for diabetic retinopathy occurence | 1 month
  obstructive sleep apnea is defined as apnea-hypopnea index > 15 on polysomnography

SECONDARY OUTCOMES:
Correlation between severity of obstructive sleep apnea and presence of diabetic retinopathy | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Marie Bruyneel, MD, PhD, Principal Investigator — Centre hospitalier universitaire St Pièrre - Pneumologie/Labo du sommeil
Locations (1):
- Centre Hospitalier Universitaire Saint Pièrre, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altaf QA, Dodson P, Ali A, Raymond NT, Wharton H, Fellows H, Hampshire-Bancroft R, Shah M, Shepherd E, Miah J, Barnett AH, Tahrani AA. Obstructive Sleep Apnea and Retinopathy in Patients with Type 2 Diabetes. A Longitudinal Study. Am J Respir Crit Care Med. 2017 Oct 1;196(7):892-900. doi: 10.1164/rccm.201701-0175OC. PMID 28594570
- [Background] Mok Y, Tan CW, Wong HS, How CH, Tan KL, Hsu PP. Obstructive sleep apnoea and Type 2 diabetes mellitus: are they connected? Singapore Med J. 2017 Apr;58(4):179-183. doi: 10.11622/smedj.2017027. PMID 28429032
- [Background] Vujosevic S, Midena E. Diabetic Retinopathy in Italy: Epidemiology Data and Telemedicine Screening Programs. J Diabetes Res. 2016;2016:3627465. doi: 10.1155/2016/3627465. Epub 2016 Nov 21. PMID 27990441
- [Background] Zhou Y, Zhang Y, Shi K, Wang C. Body mass index and risk of diabetic retinopathy: A meta-analysis and systematic review. Medicine (Baltimore). 2017 Jun;96(22):e6754. doi: 10.1097/MD.0000000000006754. PMID 28562529